CLINICAL TRIAL: NCT01133327
Title: Adapt™ Monorail™ Carotid Stent System: A Postmarket Clinical Follow-up Study
Brief Title: Adapt Monorail Carotid Stent System: A Postmarket Clinical Follow-up Study
Acronym: ASTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: CRO genae (Unknown); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTI
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Carotid Artery Disease; Carotid Stenosis; Stroke
Keywords: Carotid Artery Stenting; High Risk patient; Carotid artery stenosis; stroke; Carotid artery disease; ASTI study; Adapt Carotid Stent system; FilterWire EZ Embolic Protection System
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adapt Carotid Stent System (Experimental): Intervention with Adapt Carotid Stent System with the FilterWire EZ System
  Interventions: Device: Carotid Artery Stenting

INTERVENTIONS:
Device: Carotid Artery Stenting — The Adapt Carotid Stent System is intended to deliver a self-expanding Stent to the extra-cranial carotid arteries via a sheathed percutaneous Monorail delivery system. The Adapt Carotid Stent is a closed cell, self-expanding, rolled nitinol (nickel-titanium alloy) sheet. The stent is thin, flexible and expands to appose the vessel wall.
  The FilterWire EZ System is a temporary intravascular guide wire filtration system that is placed in the vessel distal to the lesion to be treated. It consists of either a polyurethane filter bag 1.5 cm in length or a Bionate (polycarbonate urethane) filter bag, 1.0 cm in length attached near the distal end of a 0.014" silicone coated stainless steel guide wire by means of a collapsible, self-conforming, Nitinol filter loop wire.
  Other Names: Adapt Monorail Carotid Stent system 21mm, 32mm, 40mm; FilterWire Embolic Protection System 3.5 mm - 5.5 mm

SUMMARY:
The purpose of this study is to get outcomes data for the Adapt Monorail Carotid System used in conjunction with the FilterWire Embolic protection system for treatment of patients that suffer from carotid artery stenosis and that cannot have surgery due to high risk factors.

DETAILED DESCRIPTION:
According to the World Health Organization, 15 million people suffer stroke each year. Of these, 5 million die and another 5 million are permanently disabled. Predominant mechanism responsible for stroke is embolism from proximal rupture of atherosclerotic plaque and thrombus. 25-30% of stroke deaths related to the carotid stenosis. The primary therapy for carotid occlusive disease is the surgical removal of this atherosclerotic plaque from inside the artery. Another treatment option for subjects with significant surgical risk factors has been found: the carotid artery stenting is a non-surgical procedure which unblocks narrowing of the carotid artery lumen by inserting a small metal tube (stent) to keep the plaque against the wall of the artery to improve blood flow.

ELIGIBILITY:
Inclusion Criteria:

* High-risk for carotid endarterectomy due to anatomical or co-morbid conditions and either has neurological symptoms and ≥ 50% stenosis, via angiography or is asymptomatic and has ≥ 80% stenosis, via angiography
* Target lesion located in the common carotid artery (CCA), internal carotid artery (ICA), or carotid bifurcation
* Arterial segment to be stented has a diameter between 4mm and 9mm
* Age ≥ 18 years
* Life expectancy > 12 months from the date of the index procedure

Exclusion Criteria:

* Contraindication to percutaneous transluminal angioplasty (PTA)
* Severe vascular tortuosity or anatomy that would preclude the safe introduction of a guide catheter, sheath, embolic protection system or stent system
* Lesions in the ostium of the common carotid artery
* Occlusion of the target vessel
* Evidence of intraluminal thrombus
* Known sensitivity to nickel-titanium
* Known allergy to heparin, aspirin or other anticoagulant/ antiplatelet therapies, or is unable or unwilling to tolerate such therapies
* Uncorrectable bleeding disorders, or will refuse blood transfusions
* History of prior life-threatening contrast media reaction
* Previous stent placement in the target vessel
* Evolving stroke or intracranial hemorrhage
* Previous intracranial hemorrhage or brain surgery within the past 12 months
* Clinical condition that makes endovascular therapy impossible or hazardous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
30-day rate of major adverse events | 30-day postprocedure
  30-day rate of major adverse events, defined as the cumulative incidence of any peri-procedural (less or equal to 30 days postprocedure) death, stroke, or Myocardial Infarction

SECONDARY OUTCOMES:
Late ipsilateral stroke | 31 through 365 days post procedure
System Technical Success | the procedure time
  successful placement and retireval of the FilterWire EZ System, and the successful deployment of the Adapt Carotid Stent sytem in the target carotid artery, with a residual stenosis < or equal to 30% as determined by the core lab.
Device Malfunctions | from index procedure to 365 days post procedure
  Define as any failure of the device to meet performance specifications or otherwise perform as intended, as defined by the investigator.
Serious device-related and procedure-device related Events | from index procedure to 365 days post procedure
Target Lesion Revascularization | from end of index procedure to 365 days postprocedure
  any surgical or percutaneous attempt to revascularize the target lesion after the initial or index treatment when the diameter restenosis is either equal to 50% or above with symptoms related to the target lesion or 80% or above without symptoms related to the target lesion.
In-stent Restenosis | from end of index procedure to 365 days post procedure
Major Adverse Events Rate by subgroups | from index procedure to 365 days post procedure
  Major Adverse Events Rate by subgroups
  * symptomatic and asymptomatic status
  * per center

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator; Monika Hanisch, PhD, Study Director — Boston Scientific Corporation
Locations (11):
- Belgium (3):
  - A.Z. Sint Blasius, Dendermonde, East-Flanders
  - Imelda Ziekenhuis, Bonheiden
  - CHU Sart Tilman, Liège
- Germany (6):
  - Königin Elisabeth Herzberge, Berlin
  - Klinikum Dortmund, Dortmund
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Park KH, Leipzig
  - Klinikum Neuperlach Munich, Munich
  - Radiologische Universitätklinik, Tübingen
- Spain (2):
  - Hospital Juan Canalejo, A Coruña
  - Complejo Hospitalario de Toledo, Toledo

REFERENCES:
- [Background] Coward LJ, Featherstone RL, Brown MM. Safety and efficacy of endovascular treatment of carotid artery stenosis compared with carotid endarterectomy: a Cochrane systematic review of the randomized evidence. Stroke. 2005 Apr;36(4):905-11. doi: 10.1161/01.STR.0000158921.51037.64. Epub 2005 Mar 3. PMID 15746454
- [Background] Nadim Al-Murbarak et al. Carotid Artery Stenting. Lippincott Williams & Wilkins, 2004
- [Background] Hopkins LN, Myla S, Grube E, Wehman JC, Levy EI, Bersin RM, Joye JD, Allocco DJ, Kelley L, Baim DS. Carotid artery revascularization in high surgical risk patients with the NexStent and the Filterwire EX/EZ: 1-year results in the CABERNET trial. Catheter Cardiovasc Interv. 2008 Jun 1;71(7):950-60. doi: 10.1002/ccd.21564. PMID 18412236
- [Background] World Health Report - 2007, from the World Health Organization. Accesses October 31, 2009
- [Background] Stroke Facts and Statistics from the Center of Disease Control and Prevention,Division for Heart Disease and Stroke Prevention. Available at http://www.cdc.gov/Stroke/stroke_facts.htm. Page last modified February 12, 2009. Accessed October 23, 2009.
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] National Institute of Heath / National Institute of Neurological Disorders and Stroke. NIH Stroke Scale. Available at http://www.ninds.nih.gov/doctors/NIH_Stroke_Scale_Booklet.pdf. Accessed October 23, 2009.